CLINICAL TRIAL: NCT04901468
Title: A-EYE: A Mixed Quantitative and Qualitative Study to Develop and Evaluate the Application of Artificial Intelligence (AI) Methods Using Retinal Imaging for the Identification of Adverse Retinal Changes Associated With Cancer Therapies.
Acronym: A-EYE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Principal Investigator, Tariq Aslam, Professor Of Ophthalmology and Interface Technologies and Consultant Ophthalmologist, University of Manchester
Other Study IDs: NHS001768
Record Dates: First submitted 2021-05-17; First posted 2021-05-25 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: All Comers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — This is an observational study

SUMMARY:
This is a data collection study involving the gathering of clinical data and OCT (optical coherence tomography) scans from 350 patients.

The purpose of this study is to gather data to help develop an AI algorithm to detect eye abnormalities specifically those related to certain cancer treatments.

At the end of the study interviews will be held with expert ophthalmologists to assess the acceptability of implementing AI into clinical practice.

DETAILED DESCRIPTION:
Many cancer patients will access new treatments through clinical trials. These treatments have often never been tested in humans and therefore, are likely to have unknown side effects. Some of these side effects include changes to the eye, such as blindness.

Ahead of patients taking part in these trials there is often little planning done to manage potential side effects on the eye. Additionally, accessing the expertise of eye specialists is not always available and often referral to a specialist is only given when eye symptoms have become advanced. These delays in identifying side effects on the eye also delays treatment and follow-up management. Providing patients access to this expertise would help in the detection and management of treatment side effects, however, due to demands on resources this access is not always readily available.

The aim of this study is to create an artificial intelligence (AI) program that can detect changes to the eye related to disease, which, in the future, can be specifically used in cancer patient care. Additionally, developing an AI program to detect cancer related side effects to the eye will go a significant way in easing the burden on the health care system and improve side effects from new cancer treatments.

This study will involve the collection of eye scans and medical data from participants at the Manchester Royal Eye Hospital. These will then be used to develop AI methods to detect changes in the eye related to those seen by patients on cancer treatment. The AI will then be compared with the assessments of eye specialists to assess if they give similar results.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for the study if all inclusion criteria are met:

1. Voluntary informed consent.
2. Aged at least 18 years.
3. Fully registered patient attending the Manchester Royal Eye Hospital
4. Patients are having an optical diagnostic imaging as part of their standard of care.

Exclusion Criteria:

Patients are excluded from the study if any of the following criteria apply:

1. Patient who are deemed clinically unable to be scanned by healthcare professional.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients at the Manchester Royal Eye Hospital who meet the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure of the diagnostic accuracy of the AI algorithm against gold standard clinical assessment associated with cancer treatment. | 12 months

SECONDARY OUTCOMES:
Sensitivity of the AI in identifying clinically relevant lesions as defined by an ophthalmologist. Specificity of the AI in identifying clinically relevant lesions as defined by an ophthalmologist. | 12 months

OTHER OUTCOMES:
F1 score of the proposed algorithm compared against baseline algorithms. | 13 months
Recorded questionnaire/ interview with ophthalmologist and cancer specialists. | 9 months
Number of novel relationships identified | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Royal Eye Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No